CLINICAL TRIAL: NCT01037413
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, WITHIN-SUBJECT CONTROLLED STUDY TO EVALUATE EFFICACY AND SAFETY OF EXC 001 FOR THE AMELIORATION OF SCARRING FOLLOWING REVISION OF SCARS RESULTING FROM PRIOR BREAST SURGERY IN ADULT FEMALE SUBJECTS
Brief Title: Safety and Efficacy Study of EXC 001 to Improve the Appearance of Scars From Prior Breast Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: EXC 001-203; B5301011 (Other: Alias Study Number)
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Scar Prevention
Keywords: Scarring; Cicatrix; Fibrosis; Pathologic Process
MeSH Terms: conditions — Cicatrix; Fibrosis; Pathologic Processes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EXC 001 (Experimental)
  Interventions: Drug: EXC 001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EXC 001 — Multiple intradermal injections of EXC 001 and placebo
  Arms: EXC 001
Drug: Placebo — Multiple intradermal injections of EXC 001 and placebo
  Arms: Placebo

SUMMARY:
This study will compare how well EXC 001 works to improve the appearance of scars in subjects undergoing breast scar revision surgery. The study will also evaluate the safety of EXC 001 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have previously had breast surgery resulting in unacceptable scars
* Subject has chosen to have the breast scars revised
* Subjects must not be pregnant or lactating

Exclusion Criteria:

* Currently pregnant or pregnant during the 6 months prior to inclusion in the study, or lactating
* Participation in another clinical trial within 30 days prior to the start of the study
* Any other condition or prior therapy, which, in the opinion of the PI, would make the subject unsuitable for this study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2009-12-22 (Actual); Primary Completion 2010-04-09 (Actual); Study Completion 2010-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Scripps medical, La Jolla, California
  - Northwestern University,Division of Plastic Surgery, Chicago, Illinois
  - Body Aesthetic Plastic Surgery, St Louis, Missouri
  - Jewell Plastic Surgery Center, Eugene, Oregon
  - Connall Consmetic Surgery, Tualatin, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EXC001-203&StudyName=Safety%20and%20Efficacy%20Study%20of%20EXC%20001%20to%20Improve%20the%20Appearance%20of%20Scars%20From%20Prior%20Breast%20Surgery%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who elected to revise appearance of bilateral scars from previous breast surgery, were recruited in this study. Study had 2 parts- Part A and B. Participants with negative skin sensitization in Part A (skin testing) were assigned to Part B (scar revision surgery) of the study.
Pre-assignment Details: Safety assessment was not planned separately for EXC 001 (PF-0647387) and placebo. All participants acted as their own control receiving both EXC 001 and placebo on the same days during Part B of the study.
Groups:
- EXC 001 During Part A: In Part A, participants received 2 intradermal injections of EXC 001 at a dose of 5 milligram (mg) on Day 1 and 21, on lower back. Third 5 mg intradermal injection of EXC 001 was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to scar revision surgery.
- EXC 001 + Placebo During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent scar revision surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear centimeter (cm) to a 6 cm section of both sides of scar on one breast and 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of scar on another breast (other breast than which received EXC 001), at Week 2, 5, 8, and 11 after the surgical incision was closed.
Period: Part A: Skin Testing
Arm/Group | EXC 001 During Part A | EXC 001 + Placebo During Part B
Started | 25 | 0
Completed | 23 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Part B: Scar Revision
Arm/Group | EXC 001 During Part A | EXC 001 + Placebo During Part B
Started | 0 (Participants who tested negative for skin sensitization proceeded to Part B of the study. .) | 23 (Participants who completed Part A of the study and were negative for skin sensitization.)
Treated | 0 | 22
Completed | 0 | 21
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Assigned But Not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Groups:
- All Enrolled Participants: All participants who were enrolled in the study.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Expert Panel Scar Assessment Score at Week 12
Description: Scar assessment by an expert panel was done on blinded photographs using 100 millimeter (mm) visual analog scale (VAS) where a score of 0 mm = best possible scar and a score of 100 mm = worst possible scar, where higher scores indicate worse condition.
Time Frame: Part B: Week 12
Population: Completer population included all participants who had missed not more than 1 dose of study drug, had the Week 12 assessment and non-missing data for VAS scar assessment score.
Measure: Mean (Standard Deviation); unit: millimeter
Groups:
- EXC 001 During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent scar revision surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of scar on one breast at Week 2, 5, 8, and 11 after the surgical incision was closed.
- Placebo During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent scar revision surgery on Day 1 and then received 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of scar on another breast (other breast than which received EXC 001), at Week 2, 5, 8, and 11 after the surgical incision was closed.
Arm/Group | EXC 001 During Part B | Placebo During Part B
Number analyzed (Participants) | 21 | 21
millimeter | 36.6 (12.68) | 51.4 (14.54)
Statistical Analysis 1: Comparison: EXC 001 During Part B vs Placebo During Part B; Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -14.7, 95% CI 2-sided [-21.3 to -8.1]

2. Secondary Outcome: Expert Panel Scar Assessment Score at Week 8 and 24
Description: Scar assessment by an expert panel was done on blinded photographs using 100 mm VAS where a score of 0 mm = best possible scar and a score of 100 mm = worst possible scar, where higher scores indicate worse condition.
Time Frame: Part B: Week 8 and 24
Population: Completer population included all participants who had missed not more than 1 dose of study drug, had the Week 12 assessment and non-missing data for VAS scar assessment score. Here 'Number Analyzed' signifies those participants who were evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | EXC 001 During Part B | Placebo During Part B
Number analyzed (Participants) | 21 | 21
millimeter
  Week 8: number analyzed (Participants) | 19 | 19
  Week 8 | 34.7 (11.18) | 49.4 (13.96)
  Week 24 | 30.7 (13.55) | 56.7 (22.56)
Statistical Analysis 1: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 8: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -14.8, 95% CI 2-sided [-21.2 to -8.3]
Statistical Analysis 2: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -26.0, 95% CI 2-sided [-34.3 to -17.7]

3. Secondary Outcome: Physician Observer Scar Assessment Score at Week 12 and 24
Description: Physician observer assessment of scar was done using a valid published 10-point rating scale. Physician rated vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion for a scar on a score of 1= normal skin to 10= worst scar imaginable, where higher scores indicate worse condition. Composite score was the sum of all the scores except the overall opinion score and range from 6 (best score) to 60 (worst score), where higher scores indicate worse condition.
Time Frame: Part B: Week 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 During Part B | Placebo During Part B
Number analyzed (Participants) | 21 | 21
units on a scale
  Week 12: Vascularity | 4.0 (1.75) | 5.2 (1.67)
  Week 12: Pigmentation | 3.4 (1.33) | 4.6 (1.80)
  Week 12: Thickness | 3.8 (1.58) | 5.4 (2.18)
  Week 12: Relief | 3.4 (1.69) | 5.2 (2.47)
  Week 12: Pliability | 3.6 (1.66) | 4.7 (2.15)
  Week 12: Surface Area | 3.9 (1.53) | 5.3 (1.77)
  Week 12: Overall Opinion | 3.7 (1.46) | 5.5 (1.83)
  Week 12: Composite Score | 22.1 (7.53) | 30.5 (10.42)
  Week 24: Vascularity | 3.5 (1.29) | 5.8 (1.95)
  Week 24: Pigmentation | 3.5 (1.21) | 5.4 (1.86)
  Week 24: Thickness | 4.0 (1.82) | 5.8 (1.83)
  Week 24: Relief | 3.2 (1.78) | 5.6 (2.29)
  Week 24: Pliability | 3.2 (1.73) | 5.2 (2.34)
  Week 24: Surface Area | 3.7 (1.71) | 5.9 (1.80)
  Week 24: Overall Opinion | 3.6 (1.43) | 6.0 (1.70)
  Week 24: Composite Score | 21.0 (7.79) | 33.6 (10.11)
Statistical Analysis 1: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Vascularity: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.033, t-test, 2 sided; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.3 to -0.1]
Statistical Analysis 2: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Pigmentation: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.9 to -0.4]
Statistical Analysis 3: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Thickness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.5 to -0.8]
Statistical Analysis 4: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Relief: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.7 to -1.0]
Statistical Analysis 5: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Pliability: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.012, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.9 to -0.3]
Statistical Analysis 6: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Surface Area: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.4 to -0.5]
Statistical Analysis 7: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Overall Opinion: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.6 to -1.1]
Statistical Analysis 8: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -8.4, 95% CI 2-sided [-12.7 to -4.0]
Statistical Analysis 9: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Vascularity: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.2 to -1.4]
Statistical Analysis 10: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Pigmentation: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.9 to -0.9]
Statistical Analysis 11: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Thickness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.8 to -0.8]
Statistical Analysis 12: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Relief: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-3.6 to -1.3]
Statistical Analysis 13: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Pliability: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.005, t-test, 2 sided; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.2 to -0.7]
Statistical Analysis 14: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Surface Area: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.1 to -1.2]
Statistical Analysis 15: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Overall Opinion: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-3.3 to -1.5]
Statistical Analysis 16: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -12.6, 95% CI 2-sided [-17.7 to -7.4]

4. Secondary Outcome: Participant Observer Scar Assessment Score at Week 12 and 24
Description: Participants rated pain, itching, color, stiffness, thickness, irregularity, and overall opinion of scar on 10-point scale. For pain and itching associated with scar: range =1 (no, not at all) to 10 (yes, worst imaginable) and for other parameters associated with scar compared to normal skin: range =1 (no, same as normal skin) to 10 (yes, very different), where higher scores indicate worse condition. Composite score = sum of all scores except overall opinion, range 6 (best) to 60 (worst), where higher scores indicate worse condition. Scar appearance composite score = sum of all scores except overall opinion, pain and itching, range 4 (best) to 40 (worst), where higher scores indicate worse condition.
Time Frame: Part B: Week 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 During Part B | Placebo During Part B
Number analyzed (Participants) | 21 | 21
units on a scale
  Week 12: Pain | 2.0 (2.13) | 2.7 (1.93)
  Week 12: Itching | 2.6 (2.82) | 3.0 (2.87)
  Week 12: Color | 6.3 (3.07) | 6.8 (2.91)
  Week 12: Stiffness | 4.0 (2.81) | 5.1 (3.42)
  Week 12: Thickness | 4.4 (2.94) | 5.5 (2.96)
  Week 12: Irregular | 4.6 (3.23) | 5.8 (3.11)
  Week 12: Overall Opinion | 3.7 (1.90) | 4.8 (2.62)
  Week 12: Composite Score | 24.0 (13.46) | 28.9 (13.79)
  Week 12: Scar Appearance Composite Score | 19.3 (10.95) | 23.3 (10.97)
  Week 24: Pain | 1.5 (1.08) | 2.4 (2.36)
  Week 24: Itching | 1.9 (2.00) | 2.5 (2.32)
  Week 24: Color | 5.2 (3.14) | 7.0 (2.77)
  Week 24: Stiffness | 3.6 (2.62) | 5.8 (3.33)
  Week 24: Thickness | 3.6 (2.48) | 6.0 (3.26)
  Week 24: Irregular | 4.3 (2.49) | 6.1 (3.20)
  Week 24: Overall Opinion | 4.1 (2.48) | 6.5 (2.93)
  Week 24: Composite Score | 20.1 (9.96) | 29.9 (13.80)
  Week 24: Scar Appearance Composite Score | 16.7 (9.37) | 24.9 (11.61)
Statistical Analysis 1: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12 Pain: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.067, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.3 to 0.0]
Statistical Analysis 2: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Itching: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.413, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.2 to 0.5]
Statistical Analysis 3: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Color: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.401, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.6 to 0.7]
Statistical Analysis 4: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Stiffness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.083, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.4 to 0.2]
Statistical Analysis 5: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Thickness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.052, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.3 to 0.0]
Statistical Analysis 6: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Irregular: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.036, t-test, 2 sided; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.3 to -0.1]
Statistical Analysis 7: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Overall Opinion: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.045, t-test, 2 sided; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.1 to -0.0]
Statistical Analysis 8: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.054, t-test, 2 sided; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-9.9 to 0.1]
Statistical Analysis 9: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 12, Scar Appearance Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.065, t-test, 2 sided; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-8.2 to 0.3]
Statistical Analysis 10: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Pain: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.079, t-test, 2 sided; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.0 to 0.1]
Statistical Analysis 11: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Itching: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.158, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.5 to 0.3]
Statistical Analysis 12: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Color: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.010, t-test, 2 sided; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.0 to -0.5]
Statistical Analysis 13: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Stiffness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-3.5 to -0.8]
Statistical Analysis 14: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Thickness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.005, t-test, 2 sided; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.0 to -0.8]
Statistical Analysis 15: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Irregular: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.032, t-test, 2 sided; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.5 to -0.2]
Statistical Analysis 16: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Overall Opinion: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.8 to -0.9]
Statistical Analysis 17: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.006, t-test, 2 sided; Mean Difference (Final Values) = -9.8, 95% CI 2-sided [-16.4 to -3.1]
Statistical Analysis 18: Comparison: EXC 001 During Part B vs Placebo During Part B; Week 24, Scar Appearance Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.004, t-test, 2 sided; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-13.4 to -3.0]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included SAEs and all non-SAEs that occurred during the study.
Time Frame: Part A: Day 1; Part B, Active Dosing: Week 2 up to Week 13; Part B, Post Dosing: Week 13 to end of the study (Week 24)
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- EXC 001 During Part A: In Part A, participants received 2 intradermal injections of EXC 001 at a dose of 5 mg on Day 1 and 21, on lower back. Third 5 mg intradermal injection of EXC 001 was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to scar revision surgery.
- EXC 001 + Placebo During Part B, Active Dosing Phase: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent scar revision surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of scar on one breast and 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of scar on another breast (other breast than which received EXC 001), at Week 2, 5, 8, and 11 after the surgical incision was closed. Active dosing was the time period from Week 2 to Week 13.
- Part B, Post Dosing Phase: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants who received treatment in active dosing phase were followed up from Week 13 until end of the study in post dosing phase.
Arm/Group | EXC 001 During Part A | EXC 001 + Placebo During Part B, Active Dosing Phase | Part B, Post Dosing Phase
Number analyzed (Participants) | 25 | 22 | 22
Participants
  AEs | 9 | 16 | 3
  SAEs | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included the assessment of skin; head, ears, eyes, nose, and throat; respiratory; cardiovascular; abdomen; musculoskeletal; neurological; gastrointestinal; genitourinary; endocrine and lymph nodes. Abnormal physical examination findings was based on investigator's discretion.
Time Frame: Screening (up to Day 21 prior to Day 1 of Part A), Part B: Day 1, Week 12
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug. Here, "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: In Part A, participants received 2 intradermal injections of EXC 001 at a dose of 5 mg on Day 1 and 21, on lower back. Third 5 mg intradermal injection of EXC 001 was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery. Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent scar revision surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of scar on one breast and 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of scar on another breast, at Week 2, 5, 8, and 11 after the surgical incision was closed.
Arm/Group | Overall Study
Number analyzed (Participants) | 25
Participants
  Screening | 14
  Day 1 of Part B: number analyzed (Participants) | 22
  Day 1 of Part B | 3
  Week 12 of Part B: number analyzed (Participants) | 22
  Week 12 of Part B | 1

7. Secondary Outcome: Number of Participants With Clinically Significant Findings in Electrocardiogram (ECG)
Description: Number of participants with clinically significant abnormality in ECG were reported. Clinical significance was based on investigator's discretion.
Time Frame: Screening (up to Day 21 prior to Day 1 of Part A), Part B: Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 25
Participants
  Screening | 0
  Part B: Week 12: number analyzed (Participants) | 22
  Part B: Week 12 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Findings in Laboratory Examinations
Description: Laboratory analysis included hematology, biochemistry and urinalysis. Hematology range: basophils (bas) 0-0.2, eosinophils (eos) 0-0.4, leukocytes (leu) 4-10.5, lymphocytes (lym) 0.7-4.5, neutrophils (neu) 1.8-7.8, platelet 140-415, monocytes (mon) 0.1-1 in 10^9 per liter; bas/leu 0-3, eos/leu 0-7, lym/leu 14-46, mon/leu 4-13, neu/leu and neu/leu 40-74 in percentage, erythrocytes 3.8-5.1 10^12/L, hematocrit 0.34-0.44 L/L, hemoglobin 115-150 gram per liter (g/L). Biochemistry range: creatine kinase 24-173, alkaline phosphatase 25-150, alanine aminotransferase (AT) and aspartate AT 0-40 in International units per liter; creatinine 50-88, urate 89-399, bilirubin 2-21 in micromole per liter, glucose 3.6-5.5, potassium 3.5-5.5, sodium 135-148, blood urea nitrogen 1.8-9.3 in millimole/L, albumin 35-55 g/L. Urinalysis parameters: pH (5-7.5), specific gravity (1.005-1.03). Participants with clinically significant findings were reported.
Time Frame: Screening (up to Day 21 prior to Day 1 of Part A), Part B: Day 1 up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: In Part A, participants received 2 intradermal injections of EXC 001 at a dose of 5 milligram (mg) on Day 1 and 21, on lower back. Third 5 mg intradermal injection of EXC 001 was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery. The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until the day of surgery in Part B. Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent scar revision surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of scar on one breast and 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of scar on another breast, at Week 2, 5, 8, and 11 after the surgical incision was closed.
Arm/Group | Overall Study
Number analyzed (Participants) | 25
Participants
  Screening | 0
  Part B: Day 1 up to Week 12: number analyzed (Participants) | 22
  Part B: Day 1 up to Week 12 | 2

9. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs
Description: Following vital sign parameters were assessed: diastolic blood pressure, systolic blood pressure, respiration rate, pulse rate, and temperature. Clinical significance was based on investigator's discretion.
Time Frame: Screening (up to Day 21 prior to Day 1 of Part A), Part B: Day 1 up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 25
Participants
  Screening | 0
  Part B: Day 1 up to Week 12: number analyzed (Participants) | 22
  Part B: Day 1 up to Week 12 | 1

10. Secondary Outcome: Number of Participants With Positive Skin Sensitivity Reaction
Description: Participants were instructed to inform the investigator in case of any itching, redness, pain or any other symptom that appears to be a rash at the injection sites. Erythematous, raised (indurated) and edematous reactions were considered as positive skin sensitivity reactions.
Time Frame: Part A: Day 1, Part B: Week 2 up to Week 24
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- EXC 001 + Placebo During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent scar revision surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of scar on one breast and 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of scar on another breast (other breast than which received EXC 001), at Week 2, 5, 8, and 11 after the surgical incision was closed.
Arm/Group | EXC 001 During Part A | EXC 001 + Placebo During Part B
Number analyzed (Participants) | 25 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug. Safety assessment was not planned and reported separately for EXC 001 and placebo.
Groups:
- EXC 001 + Placebo During Part B, Active Dosing Phase: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent scar revision surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of scar on one breast and 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of scar on another breast (other breast than which received EXC 001), at Week 2, 5, 8, and 11 after the surgical incision was closed.
Arm/Group | EXC 001 During Part A | EXC 001 + Placebo During Part B, Active Dosing Phase | Part B, Post Dosing Phase
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 9/25 | 16/22 | 3/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXC 001 During Part A (N=25) | EXC 001 + Placebo During Part B, Active Dosing Phase (N=22) | Part B, Post Dosing Phase (N=22)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXC 001 During Part A (N=25) | EXC 001 + Placebo During Part B, Active Dosing Phase (N=22) | Part B, Post Dosing Phase (N=22)
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site oedema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Suture rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Itching scar (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Application site erythema (General disorders) | 0 | 1 | 0
Application site pruritus (General disorders) | 0 | 1 | 0
Application site scab (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Injection site exfoliation (General disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.